CLINICAL TRIAL: NCT02796144
Title: Metformin and Lorcaserin for Weight Loss in Schizophrenia
Acronym: MELT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The FDA advised of a possible health risk associated with lorcaserin and the drug is being withdrawn.
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Columbia University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-1998; 1R01DK105526-01A1 (NIH)
Record Dates: First submitted 2016-06-06; First posted 2016-06-10 (Estimated); Results first posted 2021-02-05 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2020-05

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Overweight
Keywords: schizophrenia; schizoaffective disorder; overweight; obesity; weight loss; metformin; lorcaserin
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Overweight; Obesity; Weight Loss | interventions — lorcaserin; Metformin; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lorcaserin and Metformin (Active Comparator): Lorcaserin will be administered in dosages of 10 mg with a maximum dose of 20 mg.
  Metformin will be administered in dosages of 500 mg with a maximum dose of 2,000 mg.
  Interventions: Drug: Lorcaserin; Drug: Metformin
- Lorcaserin (Active Comparator): Lorcaserin will be administered in dosages of 10 mg with a maximum dose of 20 mg.
  Interventions: Drug: Lorcaserin
- Placebo (Placebo Comparator): Matching placebos will be administered for each active drug.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lorcaserin — Max dose of 10 mg BID
  Other Names: Belviq
  Arms: Lorcaserin; Lorcaserin and Metformin
Drug: Metformin — Max dose of 1,000 mg BID
  Other Names: Glumetza, Riomet, Glucophage, and Fortamet
  Arms: Lorcaserin and Metformin
Drug: Placebo — Matching placebos will be administered for each drug.
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
Purpose: The purpose of this study is to test new pharmacologic strategies for weight loss in patients with schizophrenia, a population for which no current weight-loss treatments have gained widespread use. The goal is to recruit overweight people with schizophrenia to participate in a 52-week double-blind, randomized study to assess the efficacy and safety of lorcaserin/metformin combination treatment, lorcaserin monotherapy, and placebo on weight, body composition, and measures of glucose and lipid metabolism.

Participants: Approximately 110 subjects will be enrolled at four clinical sites (UNC Chapel Hill, Carolina Behavioral Care, Columbia University, and Augusta University)

Procedures (methods): Behavioral: All participants will be offered a behavioral intervention of weekly diet and exercise counseling aimed at modifying cardiovascular risk factors. This intervention will be provided at all in-person study visits after the Baseline Visit and supplemented with weekly interim phone calls to reinforce lessons between visits. Pharmacological Intervention: All participants who meet entry criteria will be randomized to one of the three treatment groups (lorcaserin/metformin, lorcaserin, and placebo).

DETAILED DESCRIPTION:
Overview of Procedures: All procedures will be conducted at either the UNC Hospitals outpatient clinic in Chapel Hill, NC, at the outpatient North Carolina Psychiatric Research Center (NCPRC), a specialized program of the University of North Carolina Center for Excellence in Community Mental Health in Raleigh, NC, at Carolina Behavioral Care in Hillsborough, NC, at the Lieber Schizophrenia Research Clinic at the New York State Psychiatric Institute (NYSPI) in New York, NY, or at Augusta University in Augusta, GA.

Screening: During the initial clinic visit and after giving informed consent, prospective subjects' psychiatric and medical histories will be reviewed, physical exams conducted, demographics and vital signs taken, and blood and urine collected. Fasting labs will be ordered to measure metabolic parameters (lipid profile, glucose, hemoglobin A1C, insulin and lipids) as well as a complete blood count (CBC), electrolytes, liver/renal function tests, thyroid stimulating hormone (TSH), urinalysis (UA), serum pregnancy test, and urine drug screen (UDS). The Structured Clinical Interview for DSM-IV (Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition) will be administered to confirm diagnoses and the Clinical Global Impressions-Severity (CGI-S) will be used to evaluate global psychopathology.

The baseline visit will be scheduled within 28 days of the screening visit. A battery of assessments will be administered including the Clinical Global Impressions-Severity (CGI-S), the Alcohol Use Scale (AUS), Drug Use Scale (DUS), Brief Psychiatric Rating Scale (BPRS), Columbia Suicide Severity Rating Scale (C-SSRS), three assessments to measure eating behavior (Eating Disorder Examination Questionnaire (EDE-Q), Three-Factor Eating Questionnaire (TFEQ), and Food Craving Inventory (FCI)). In addition to the paper pencil assessments, a 24 hour food recall assessment will be administered as a telephone questionnaire by trained personnel from the UNC Nutrition and Obesity Research Center. Accelerometry will also be used to estimate subjects' sedentary and active behavior. Dual-Energy X-ray Absorptiometry (DXA) will also be conducted at the baseline visit (UNC location only). Lastly, the first behavioral intervention lesson will occur at the baseline visit, providing direct lesson instruction and a diary for subjects' to take home for recording their homework and progress.

At the completion of the baseline visit, subjects who continue to meet study inclusion criteria will be randomized to one of the three treatment groups (lorcaserin & metformin, lorcaserin, and placebo). Lorcaserin will be administered in dosages of 10mg with a maximum dose of 20mg. Metformin will be administered in dosages of 500mg with a maximum dose of 2,000mg. In addition, matching placebos will be administered for each drug. Doses will be adjusted based on subject tolerability.

All participants will be offered a behavioral intervention of weekly diet and exercise counseling aimed at modifying cardiovascular risk factors including weight, activity level, blood glucose, blood pressure and lipids. This intervention will be provided by a trained clinician in individualized sessions at all study visits after the Baseline Visit and supplemented with weekly interim phone calls to reinforce lessons between visits. The intervention was adapted from a weight-reduction program developed for patients with severe mental illnesses and was used in the Metformin in the Treatment of Antipsychotic-Induced Weight Gain in Schizophrenia (METS) and the Clinical Management of Metabolic Problems in Patients with Schizophrenia: Switching to Aripiprazole versus Continued Treatment with Olanzapine, Quetiapine, or Risperidone (CAMP) trials and is therefore well known to our research group and readily implemented as part of the current proposal.

After study enrollment, subjects will be scheduled for a Week 1 and Week 2 study visit. The purpose of these visits will be to assess medication management (i.e., symptoms, adverse events/side effects, adherence, adjust dose as indicated), collect vital signs, and provide the behavioral therapy intervention. The CGI-S will be completed again at both Week 1 and Week 2, however, the BPRS and C-SSRS will be completed at Week 2 only.

The next 5 study visits will be scheduled as bi-weekly in-person visits. These visits will be similar to Week 1 and Week, 2 with the addition of the Substance Use Scale and Alcohol Use Questionnaire. After the first two behavioral intervention sessions, interim telephone calls will be made between in-person study visits to each participant to reinforce elements of the program and to answer questions.

After the Week 12 study visit, all in-person study visits will transition to monthly visits for the rest of the year. The interim telephone calls will be made bi-weekly between the in-person study visits to each participant to continue to reinforce elements of the program and to answer questions.

At Week 52, all study measures and fasting labs will be collected again.

Vital signs, adverse events, and side effects will be obtained at all in-person study visits. Monitoring labs and appetite regulating hormones will be done at Week 12, Week 24, Week 36, and Week 52.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with a diagnosis of schizophrenia or schizoaffective disorder as defined by DSM-IV-TR criteria (see Appendix 3 and Appendix 4) and confirmed by the Structured Clinical Interview for DSM-IV (SCID).
* Duration of psychotic illness must be greater than one year, as defined by having initiated antipsychotic treatment at least 1 year prior to study enrollment.
* Must be 18-65 years of age.
* Must demonstrate adequate decisional capacity to make a choice about participating in this research study and must provide written informed consent to participate.
* BMI greater than or equal to 27 kg/m^2
* Currently treated with one or a combination of two FDA-approved antipsychotic medications (typical or atypical antipsychotics) AND on that drug regimen for at least two months prior to study entry (with stable dosages for at least 1 month).
* Concomitant medications are allowed if agents and doses are unchanged for at least 1 month prior to study entry and if these medications are not among those excluded in the Exclusion Criteria.
* Women who can become pregnant must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 4 weeks after the study in such a manner that the risk of pregnancy is minimized. Acceptable methods include oral, injectable or implanted contraceptives, intrauterine devices or barrier methods such as condoms, diaphragm and spermicides. Women who can become pregnant must have a negative serum pregnancy test at the Screening Visit.

Exclusion Criteria:

* Inpatient status
* Clinical Global Impression Severity (CGI-S) score greater than or equal to 6
* Current treatment with more than 2 antipsychotics
* HbA1c greater than or equal to 6.5%
* Diagnosis of diabetes mellitus or current treatment with insulin or oral hypoglycemics
* Current or prior treatment with metformin within the past 3 months
* Current or prior treatment with lorcaserin within the past 3 months
* Current or prior treatment with a 5-HT2B agonist (e.g. cabergoline) within the past 45 days due to potential risk for heart valve defects
* Current treatment with two or more antidepressants
* Current treatment with a single antidepressant prescribed in excess of the maximum approved dose
* Current treatment with monoamine oxidase inhibitor (MAOI) class of antidepressants (isocarboxazid, phenelzine, selegiline, tranylcypromine)
* Concurrent treatment with any of the following pro-serotonergic drugs: meperidine, buspirone, dextromethorphan, triptans, tramadol, ritonavir, tryptophan, ginseng, St. John's wort
* Diagnosis of congestive heart failure
* Uncorrected thyroid disorder
* Renal impairment as evidenced by estimated glomerular filtration rate (eGFR) 50 mL/min/1.73 m^2
* Hepatic disease (ALT, AST, or GGT > 2 times upper limit of normal (ULN), total bilirubin > 1.2 times ULN)
* Metabolic acidosis (serum CO2 <20 mEq/L)
* Known hypersensitivity to metformin or lorcaserin
* Women who are pregnant or breastfeeding
* Recent (in the past 30 days) or scheduled radiological studies involving iodinated contrast material
* Alcohol abuse/dependence as determined by SCID within the past month
* Other serious and unstable medical condition in the judgment of the investigator
* DSM-IV diagnosis of mental retardation or dementia
* Any medication (prescription or non-prescription) used for weight loss must have been discontinued 3 months prior to study entry.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2016-09; Primary Completion 2020-02-14 (Actual); Study Completion 2020-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars F. Jarskog, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (4):
- United States (4):
  - Augusta University, Augusta, Georgia
  - New York State Psychiatric Institute (NYSPI), Columbia University, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Carolina Behavioral Care, Hillsborough, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brar JS, Ganguli R, Pandina G, Turkoz I, Berry S, Mahmoud R. Effects of behavioral therapy on weight loss in overweight and obese patients with schizophrenia or schizoaffective disorder. J Clin Psychiatry. 2005 Feb;66(2):205-12. doi: 10.4088/jcp.v66n0208. PMID 15705006
- [Background] Jarskog LF, Hamer RM, Catellier DJ, Stewart DD, Lavange L, Ray N, Golden LH, Lieberman JA, Stroup TS; METS Investigators. Metformin for weight loss and metabolic control in overweight outpatients with schizophrenia and schizoaffective disorder. Am J Psychiatry. 2013 Sep;170(9):1032-40. doi: 10.1176/appi.ajp.2013.12010127. PMID 23846733
- [Background] Stroup TS, McEvoy JP, Ring KD, Hamer RH, LaVange LM, Swartz MS, Rosenheck RA, Perkins DO, Nussbaum AM, Lieberman JA; Schizophrenia Trials Network. A randomized trial examining the effectiveness of switching from olanzapine, quetiapine, or risperidone to aripiprazole to reduce metabolic risk: comparison of antipsychotics for metabolic problems (CAMP). Am J Psychiatry. 2011 Sep;168(9):947-56. doi: 10.1176/appi.ajp.2011.10111609. Epub 2011 Jul 18. PMID 21768610

RESULTS

PARTICIPANT FLOW:
Groups:
- Lorcaserin and Metformin: Lorcaserin will be administered in dosages of 10 mg with a maximum dose of 20 mg.
  Metformin will be administered in dosages of 500 mg with a maximum dose of 2,000 mg.
  Lorcaserin: Max dose of 10 mg BID
  Metformin: Max dose of 1,000 mg BID
Period: Overall Study
Arm/Group | Lorcaserin and Metformin | Lorcaserin | Placebo
Started | 23 | 24 | 24
Completed | 18 | 21 | 18
Not Completed | 5 | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lorcaserin and Metformin | Lorcaserin | Placebo | Total
Number analyzed (Participants) | 23 | 24 | 24 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 22 | 24 | 24 | 70
  >=65 years | 1 | 0 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.52 (11.45) | 43.75 (10.16) | 38.25 (9.87) | 40.85 (10.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 9 | 24
  Male | 13 | 19 | 15 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 12 | 10 | 13 | 35
  White | 9 | 13 | 8 | 30
  More than one race | 1 | 1 | 1 | 3
  Unknown or Not Reported | 1 | 0 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 3 | 3 | 4 | 10
  Ethnicity: Not Hispanic or Latino | 20 | 21 | 20 | 61
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 24 | 24 | 71

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight in Participants Assigned to Lorcaserin/Metformin Combination Treatment and Placebo
Description: Change in body weight in participants assigned to lorcaserin/metformin combination treatment and participants assigned to placebo from baseline to last study visit (up to 52 weeks)
Time Frame: Baseline, Last Observed Visit (Up to 52 weeks)
Measure: Mean (Standard Error); unit: pounds
Arm/Group | Lorcaserin and Metformin | Placebo
Number analyzed (Participants) | 23 | 24
pounds | -13.05 (2.97) | -3.02 (2.29)

2. Secondary Outcome: Change in Body Weight in Participants Assigned to Lorcaserin Monotherapy Treatment and Placebo
Description: Change in body weight in participants assigned to lorcaserin monotherapy treatment and participants assigned to placebo from baseline to last study visit (up to 52 weeks)
Time Frame: Baseline, Last Observed Visit (Up to 52 weeks)
Measure: Mean (Standard Error); unit: pounds
Arm/Group | Lorcaserin | Placebo
Number analyzed (Participants) | 24 | 24
pounds | -5.18 (2.43) | -3.02 (2.29)

3. Secondary Outcome: Change in HDL Cholesterol
Description: high-density lipoprotein
Time Frame: Baseline, Last Observed Visit (Up to 52 weeks)
Population: The modified intent to treat (MITT) population included all randomized participants. Analyses using the MITT population were based on subjects with both baseline and post-treatment measures.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Lorcaserin and Metformin | Lorcaserin | Placebo
Number analyzed (Participants) | 20 | 22 | 18
mg/dL | 3.8 (1.27) | 1.45 (1.71) | -0.78 (2.63)

4. Secondary Outcome: Change in LDL Cholesterol
Description: low-density lipoprotein
Time Frame: Baseline, Last Observed Visit (Up to 52 weeks)
Population: as for outcome 3
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Lorcaserin and Metformin | Lorcaserin | Placebo
Number analyzed (Participants) | 20 | 22 | 18
mg/dL | -7.60 (3.87) | -10.86 (5.40) | -6.83 (5.03)

5. Secondary Outcome: Change in Triglycerides
Description: serum triglycerides
Time Frame: Baseline, Last Observed Visit (Up to 52 weeks)
Population: as for outcome 3
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Lorcaserin and Metformin | Lorcaserin | Placebo
Number analyzed (Participants) | 20 | 22 | 19
mg/dL | -18.60 (12.86) | -19.68 (14.97) | -3.11 (13.43)

6. Secondary Outcome: Change in Total Cholesterol
Description: Total Cholesterol
Time Frame: Baseline, Last Observed Visit (Up to 52 weeks)
Population: as for outcome 3
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Lorcaserin and Metformin | Lorcaserin | Placebo
Number analyzed (Participants) | 20 | 22 | 19
mg/dL | -9.05 (3.96) | -13.45 (7.01) | -9.21 (4.83)

7. Secondary Outcome: Change in Hemoglobin A1c
Description: glycosylated hemoglobin
Time Frame: Baseline, Last Observed Visit (Up to 52 weeks)
Population: as for outcome 3
Measure: Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Arm/Group | Lorcaserin and Metformin | Lorcaserin | Placebo
Number analyzed (Participants) | 20 | 23 | 19
percentage of glycosylated hemoglobin | -0.03 (0.05) | 0.07 (0.08) | 0.05 (0.05)

8. Secondary Outcome: Change in Fasting Glucose
Description: fasting blood glucose
Time Frame: Baseline, Last Observed Visit (Up to 52 weeks)
Population: as for outcome 3
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Lorcaserin and Metformin | Lorcaserin | Placebo
Number analyzed (Participants) | 20 | 22 | 19
mg/dL | -4.30 (3.75) | -3.27 (2.58) | 3.53 (2.11)

ADVERSE EVENTS:
Time Frame: From the time Informed Consent was signed until the last study visit, a total duration of 52 weeks after randomization.
Arm/Group | Lorcaserin and Metformin | Lorcaserin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 1/23 | 2/24 | 3/24
Other Adverse Events (participants affected / at risk) | 20/23 | 18/24 | 16/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lorcaserin and Metformin (N=23) | Lorcaserin (N=24) | Placebo (N=24)
Hospitalization due to psychosis exacerbation (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (2)
Hospitalization due to abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Important Medical Intervention due to transient suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Generalized Hives and swelling (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lorcaserin and Metformin (N=23) | Lorcaserin (N=24) | Placebo (N=24)
Nausea (Gastrointestinal disorders) | 5 | 5 | 7
Vomiting (Gastrointestinal disorders) | 5 | 4 | 6
Diarrhea (Gastrointestinal disorders) | 8 | 5 | 5
Headache (General disorders) | 11 | 10 | 8
Dizziness (General disorders) | 8 | 5 | 5
Fatigue (General disorders) | 7 | 7 | 13
Restlessness (General disorders) | 9 | 6 | 4
Muscle twitching or spasms (Musculoskeletal and connective tissue disorders) | 6 | 5 | 8
Muscle stiffness (Musculoskeletal and connective tissue disorders) | 8 | 8 | 8
Problems with coordination (Musculoskeletal and connective tissue disorders) | 5 | 2 | 5
Excess sweating (General disorders) | 5 | 2 | 3
Racing heart rate (Vascular disorders) | 5 | 4 | 5
Confusion (Psychiatric disorders) | 4 | 1 | 3
Upper Respiratory (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-20): https://cdn.clinicaltrials.gov/large-docs/44/NCT02796144/Prot_SAP_000.pdf